CLINICAL TRIAL: NCT05708105
Title: Prediction of Intraventricular Hemorrhage Using Echocardiography and Near Infrared Spectroscopy
Acronym: PIONIRS
Status: Recruiting | Type: Observational
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: London Health Sciences Centre (Other); Foothills Medical Centre (Other); Royal Alexandra Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 486734
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Intraventricular Hemorrhage of Newborn Grade 2; Intraventricular Hemorrhage of Newborn Grade 3; Intraventricular Haemorrhage Grade IV
Keywords: Near-infrared spectroscopy; Echocardiography; Head ultrasound; Preterm neonates
MeSH Terms: interventions — Caves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cerebral near-infrared spectroscopy — Continuous cerebral NIRS will be monitored using the INVOS 5100C or 7100 Cerebral Oximeter (Medtronic, Minneapolis, MN, USA), initiated as early as feasible after birth or postnatal consent and continued until 48 hours of age. Neonatal sensors applied over a light-permeable barrier will be placed on the right or left side of forehead, like the methods used in our pilot study and in line with our clinical protocol. The continuous parameters recorded for this study using cerebral NIRS will include CrSO2 and COIx.
  Other Names: NIRS
Diagnostic Test: Functional echocardiography — The first echocardiogram will be completed as soon as possible after consent and < 24 hours of age in all cases. This will be to capture markers of early low systemic blood flow and document patent ductus arteriosus and its size, as known to be associated with IVH.
  The second scan will be performed at the end of the monitoring period, between 48-60 hours of age. This scan is planned to record the change in LVO from baseline (re-perfusion), which has been postulated to relate to development of IVH.
  Other Names: Echo
Diagnostic Test: Head Ultrasound — HUS will be paired with both echocardiograms. The first HUS will document baseline IVH status (paired with the first ECHO). The final HUS will be performed between days 4-7 of age, as per the standard clinical practice by site radiology service and will be used to confirm the final IVH status.
  Other Names: HUS

SUMMARY:
Moderate-severe intraventricular hemorrhage (msIVH, Grades II-IV) is a significant neurological complication among extremely low gestational age neonates (ELGANs, <=27+6 weeks) and is associated with long-term neuro-disabilities. In Canada, msIVH affects ~25-30% of the 1300 ELGANs born annually, with little change in incidence over last decade. Typically, it occurs between days 2-7 of age, providing a finite window of opportunity. Instituting therapies at the population level, however, exposes many low-risk infants to side effects, adversely affecting risk-benefit profile and requiring large sample sizes in trials. A targeted preventative approach, though ideal, is currently challenged by our inability to reliably identify at-risk ELGANs early after birth. Near-infrared spectroscopy (NIRS) has emerged as a promising non-invasive bedside neuromonitoring tool. Pilot studies using NIRS, including ours, found lower cerebral saturations (CrSO2) and greater periods of altered cerebral autoregulation in infants who later developed msIVH. However, a systematic planned investigation is needed to establish the predictive characteristics of NIRS-derived markers, using clinically translatable methods (cumulative burden over time-period vs. single time-point values) and identify their relative performance at different time-points during transition. Further, incorporating echocardiographic (ECHO) hemodynamic markers, known to be associated with msIVH, may allow for the establishment of robust multi-model prediction models and the gain of mechanistic hemodynamic insights to inform future management. Hence, our objective is to investigate the utility of multi-modal assessment using NIRS and ECHO for early identification of ELGANs at risk of msIVH, and generate clinically applicable predictive model(s).

DETAILED DESCRIPTION:
The overall objective is to conduct a large, adequately powered prospective cohort study to investigate the utility of combined hemodynamic assessment using NIRS and ECHO for early identification of ELGANs at risk of developing moderate-severe IVH, and to establish clinically translatable prediction models.

The specific primary aim is to examine the discriminating characteristics of NIRS-derived parameters (CrSO2 and cerebral oxygenation index [COIx, values >0.5 indicate altered cerebral autoregulation]) at 12, 18, 24, 30, 36, 42 and 48 hours of age, individually and in combination, for identifying ELGANs who subsequently develop moderate-severe IVH. The postnatal age where NIRS may best identify at-risk ELGANs is unknown and identifying these infants early within 48 hours of age may maximize its impact for employing neuroprotective strategies.

The secondary aims are:

1. To examine if adding ECHO parameters of systemic blood flow (left ventricular output [LVO], superior vena cava [SVC] flow and PDA size) and patient demographics can improve the discriminating characteristics of NIRS and generate relevant clinical prediction models.
2. To gain mechanistic insights into pathophysiology of moderate-severe IVH, by examining associations between significant abnormalities on NIRS, as identified and ECHO markers which may impact cerebral perfusion and oxygen delivery (PDA and its size, LVO, right ventricular output and left ventricular ejection fraction).

This will be novel information as potential mechanisms governing low CrSO2 or altered autoregulation in ELGANs are not known and can potentially inform future clinical preventative strategies and help design interventional trials.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born <=27+6 weeks gestational age

Exclusion Criteria:

* Known genetic or congenital anomalies that are likely to affect cardiac or cerebral oxygenation measures
* Palliative care plan prior to or immediately following delivery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Preterm infants at tertiary NICU admitted to one of four study NICUs:
  * Mount Sinai Hospital, Toronto (ON)
  * The Children's Hospital at London Health Sciences Center, London (ON)
  * Foothills Medical Centre, Calgary (AB)
  * Royal Alexandra Hospital, Edmonton (AB)
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Intraventricular hemorrhage (IVH) Status | Day 4-7 clinical head ultrasound
  IVH will be classified using Volpe's classification which is also the clinical standard for IVH classification (Grade I: Blood in germinal matrix with or without IVH less than 10% of ventricular space; Grade II: IVH occupying 10-50% of ventricular space on parasagittal view; Grade III: IVH occupying >50% of ventricle with or without ventricular echo-densities; Grade IV: periventricular hemorrhagic infarction).

CONTACTS AND LOCATIONS:
Overall Officials: Poorva Deshpande, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (4):
- Canada (4):
  - Foothillls Medical Centre, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - London Health Sciences Centre, London, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No